CLINICAL TRIAL: NCT04232774
Title: Neurotronic Ablation of Arteries for the Treatment of Type 2 Diabetes Mellitus and Its Comorbidities
Acronym: NECTAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Neurotronic, Inc. (Industry)
Collaborators: Libra Medical (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PR 2010
Record Dates: First submitted 2020-01-08; First posted 2020-01-18 (Actual); Last update posted 2023-03-27 (Actual); Status verified 2023-03

CONDITIONS: Type 2 Diabetes Mellitus With Circulatory Complciation
Keywords: Denervation; T2DM; Hypertension; Obesity
MeSH Terms: conditions — Hypertension; Obesity

STUDY DESIGN:
Intervention Model Description: This is a prospective, single-center, non-randomized, open label first-in-human (FIH) study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treated by the study device (Experimental)
  Interventions: Device: The Neurotronic arterial ablation catheter

INTERVENTIONS:
Device: The Neurotronic arterial ablation catheter — a sterile, single use catheter (device) for delivering chemical agent to achieve perivascular denervation.
  Other Names: NAA

SUMMARY:
The study is to assess the safety and feasibility of chemical denervation of multiple artery beds for the treatment of Type 2 diabetes (T2DM) and its comorbidities.

DETAILED DESCRIPTION:
Diabetes mellitus is among the most prevalent chronic diseases, affecting 435 million persons as of 2015 with an annual death toll of 1.5 million, and the overwhelming majority of these have Type 2 diabetes mellitus (T2DM). Hypertension is a common comorbidity of diabetes and present in more than 50% of diabetic patients. The risk for cardiovascular disease (CVD) is four-fold higher in patients with both DM and hypertension as compared to the normotensive non-diabetic controls. Obesity, with a prevalence of over 500 million, is another common comorbidity of diabetes. These are chronic diseases associated with increased risks of cardiovascular disease, stroke, and decreased quality of life.

Neurotronic developed a novel catheter for denervation procedure. Chemical agent is delivered locally into the adventitial space and ablates the sympathetic nerve and nerve endings in the adventitial space of the target arteries.

The purpose of the study is to assess the safety and feasibility of chemical denervation of the target arteries for the treatment of Type 2 diabetes (T2DM) and its comorbidities.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 22 and ≤ 70 years at time of enrollment.
2. Diagnosed with uncontrolled T2DM with baseline.

   1. Fasting plasma glucose ≥ 155 mg/dl (8.6 mmol/l)
   2. HbA1c levels ≥ 7.5% and < 10% (58-86 mmol/mol)]
   3. On oral anti-hyperglycemic drug regimen of at least two different drug classes, and one of the two being metformin ≥ 1500 mg/day
   4. History of positive response to metformin dosage escalation, i.e., HbA1c reduction of 0.5% or more
3. Diagnosed hypertension with baseline office blood pressure of SBP of ≥ 150 mmHg and ≤ 180 mmHg and DBP ≥ 90 mmHg.
4. BMI between 27.5 and 45 kg/m2 and weight < 400lbs.
5. Vessel diameter of 3 mm to 7 mm with a minimum arterial treatable length of 20 mm.

Exclusion Criteria:

1. T1DM or poorly controlled T2DM (defined as HbA1c >10.0%).
2. Hypoglycemia unawareness or serious hypoglycemia with loss of consciousness or confusion sufficient to prevent self-treatment in last 6 months;
3. Diagnosed proliferative retinopathy or evidence of peripheral neuropathy.
4. Lack of appropriate treatment site or anatomy precluding the intervention of the target arteries.
5. History of prior target artery intervention including balloon angioplasty, stenting, etc.
6. Arterial stenosis >50% of the normal diameter segment (diameter stenosis, compared to the angiographically normal proximal or distal segment).
7. Any abnormality or disease in one or more of the target arteries that, per the physician assessment, precludes the safe insertion of the guiding catheter (including, but not limited to, artery aneurysm, excessive tortuosity, artery calcification)
8. Known or suspected secondary hypertension, such as Cushing's disease or Cushing's Syndrome, hyperaldosteronism, pheochromocytoma, thyroid and parathyroid abnormalities, history of pre-eclampsia, onset of hypertension prior to the age of 18.
9. Use of nonsteroidal anti-inflammatory drugs (NSAIDs) for two or more days per week over the month prior to enrollment.
10. Severe or unstable cardiovascular comorbidities, such as AMI or ACS, cardiac valve stenosis, pulmonary embolism, heart failure with NYHA Class III or IV, chronic atrial fibrillation, primary pulmonary hypertension, COPD.
11. Renal transplant, history of nephrectomy or single kidney, renal tumor/cancer, known non-functioning kidney, unequal renal size (>2 cm difference in renal length between kidneys associated with a chronic kidney disease or a deterioration of the kidney function), chronic renal deficiency with eGFR ≤60ml/min/1.73m2, or on chronic renal replacement therapy.
12. Liver transplant.
13. Gastrointestinal permanent anatomic alteration surgery
14. Bleeding disorders, such as bleeding diathesis, thrombocytopenia, and severe anemia.
15. Systemic infection that the investigator judges would pose unacceptable procedural risks to the subject.
16. Known hypersensitivity to contrast media, nickel and the chemical agent that cannot be adequately pre-medicated.
17. Occlusive peripheral vascular disease that would preclude percutaneous femoral access for the procedure.
18. Subject is depressed or on antidepressants.
19. Pregnancy or breastfeeding or plan to get pregnant in next 12 months.
20. Life expectancy of less than 12 months.
21. Unwilling or unable to comply with the follow-up study requirements.
22. Lacking capacity to provide informed consent.
23. Concurrent medical condition that would affect the investigator's ability to evaluate the patient's condition or could compromise patient safety.
24. Currently participation in another pre-market drug or medical device clinical study.

Ages: 22 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2019-11-04 (Actual); Primary Completion 2023-01-17 (Actual); Study Completion 2023-01-17 (Actual)

PRIMARY OUTCOMES:
Incidence of Serious Device- and Procedure-Related Complications | at 30 Days post procedure
  This composite endpoint is defined as:
  * death
  * flow-limiting dissection of the treated one or more of the arteries requiring intervention
  * perforation of the treated artery requiring intervention
  * bleeding requiring transfusion due to severe leakage at treatment site
  * severe or occlusive thrombosis of the treated artery beds
  * distal embolization of the treated artery beds

SECONDARY OUTCOMES:
Glycemic Control (1) | at baseline and at post-procedure: 2-week, 1-month, 3-month, 6-month, 12-month and 24-month follow-up visits. Also, optionally at 3-,4- and 5-year post-procedure follow-up visits.
  Improvement of HbA1c (%) will be analyzed by absolute and relative changes. Percent subjects with decrease HbA1c will also be analyzed.
Glycemic Control (2) | at baseline and at post-procedure: 2-week, 1-month, 3-month, 6-month, 12-month and 24-month follow-up visits. Also, optionally at 3-,4- and 5-year post-procedure follow-up visits.
  Improvement of fasting glucose (mg/dl) will be analyzed by absolute and relative changes. Percent subjects with decrease fasting glucose will also be analyzed.
Hypertension Control | at baseline and at post-procedure: 2-week, 1-month, 3-month, 6-month, 12-month and 24-month follow-up visits. Also, optionally at 3-,4- and 5-year post-procedure follow-up visits.
  Improvement of blood pressure (mmHg) will be analyzed by absolute and relative changes.
Weight Control (1) | at baseline and at post-procedure: 2-week, 1-month, 3-month, 6-month, 12-month and 24-month follow-up visits. Also, optionally at 3-,4- and 5-year post-procedure follow-up visits.
  The improvement of the body weight (weight in kg) will be analyzed by absolute and relative changes.
Weight Control (2) | at baseline and at post-procedure: 2-week, 1-month, 3-month, 6-month, 12-month and 24-month follow-up visits. Also, optionally at 3-,4- and 5-year post-procedure follow-up visits.
  The improvement of the body weight will be analyzed by Body Mass Index (BMI in kg/m^2) absolute and relative changes.
Device Success | during procedure or immediately after procedure
  Device success, defined as successful introduction of the catheter, navigation to the treatment site, deployment of the features, and infusion of the chemical agent to the intended area without device malfunction that requiring abort the procedure.
Procedure Success | during procedure or immediately after procedure
  Procedure success, defined as device success without any serious device- and procedure-related complications during the procedure and prior to hospital discharge.

CONTACTS AND LOCATIONS:
Overall Officials: John Chen, Study Director — Neurotronic, Inc.
Locations (1):
- Sanatorio Italiano - Centro de Intervenciones Endovasculares, Asunción, Paraguay

IPD SHARING:
Plan to Share IPD: No